CLINICAL TRIAL: NCT07367646
Title: Development and Validation of a Multidimensional Screening Tool for Work-Related Musculoskeletal Disorders: A COSMIN-Guided Psychometric Study
Brief Title: Development of Multidimensional Screening Tool for WMSDs
Status: Not yet recruiting | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Kibum Jung, Ph.D. Candidate, Sahmyook University
Other Study IDs: SYU 2025-12-018-001
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Work-Related Musculoskeletal Disorders; Musculoskeletal Diseases; Occupational Diseases
Keywords: WMSDs; Musculoskeletal Pain; Screening Tool; Psychometrics; Occupational Health
MeSH Terms: conditions — Musculoskeletal Diseases; Occupational Diseases; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bio-pharmaceutical Industry Workers: Workers currently employed at Samsung Biologics, including both office and production staff, who meet the inclusion criteria for musculoskeletal symptoms.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Participants will complete the newly developed multidimensional screening tool and standard validation questionnaires (e.g., OSPRO-YF, FABQ, TSK) to assess musculoskeletal symptoms and psychosocial factors.

SUMMARY:
The purpose of this study is to develop a multidimensional screening tool for Work-Related Musculoskeletal Disorders (WMSDs) and to evaluate its psychometric properties. The study involves a cross-sectional survey of approximately 250 workers in the bio-pharmaceutical industry to assess the tool's structural validity, internal consistency, construct validity, and measurement invariance following COSMIN guidelines.

DETAILED DESCRIPTION:
Work-related musculoskeletal disorders (WMSDs) are a major occupational health issue. While various screening tools exist, few comprehensively assess red flags (signs of serious pathology), yellow flags (psychosocial risk factors), and physical symptoms specifically for industrial workers. This study aims to address this gap by developing a new screening tool and validating its reliability and validity. The study design follows the COSMIN (COnsensus-based Standards for the selection of health Measurement INstruments) checklist. The validation process involves a cross-sectional survey targeting 250 workers, including both office and production staff. The developed tool is designed to screen for serious medical conditions (Red flags) requiring referral, as well as to assess physical symptoms and psychosocial barriers (Yellow flags). Psychometric evaluation will specifically focus on the physical and psychosocial domains, as Red flags are typically binary screening items. Key psychometric properties to be evaluated include: 1. Structural Validity: Confirmatory Factor Analysis (CFA) will be conducted to verify the factor structure of the physical and psychosocial domains. 2. Internal Consistency: Cronbach's alpha coefficients will be calculated for these subscales. 3. Measurement Invariance: Multi-group CFA will be performed to ensure the tool functions equivalently across different job types (office vs. production). 4. Construct Validity: Correlations with established instruments (e.g., OSPRO-YF, FABQ, TSK) will be analyzed. The ultimate goal is to provide a practical and scientifically validated instrument for the early detection, triage, and management of WMSDs in workplace settings. 5. Cut-off Determination: ROC analysis will be conducted to establish optimal cut-off scores for identifying high-risk groups (Yellow flags), using established tools as a reference.

ELIGIBILITY:
Inclusion Criteria:

* Current regular employees working at the study site.
* Adults aged 19 years or older who understand the study purpose and procedures and voluntarily agree to participate in writing.
* Participants capable of reading, understanding, and self-responding to the questionnaire.
* Individuals with musculoskeletal symptoms according to NIOSH standards: symptoms lasting more than one week OR recurring at least once a month in the past 12 months (symptoms include pain, aching, stiffness, burning sensation, tingling, or numbness).

Exclusion Criteria:

* Individuals with cognitive or mental impairments that make it difficult to understand the study or complete the survey.
* Individuals suspected of having a medical emergency or severe disease requiring immediate medical attention.
* Individuals deemed unsuitable for participation by the researcher.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of workers currently employed at a bio-pharmaceutical company (Samsung Biologics) in South Korea. This includes both office workers engaged in VDT tasks and production workers involved in physical tasks who report musculoskeletal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural Validity | Baseline
  Evaluated using Confirmatory Factor Analysis (CFA). Model fit will be assessed based on stricter criteria: CFI ≥ 0.95, TLI ≥ 0.95, RMSEA ≤ 0.06, and SRMR ≤ 0.08 (Hu & Bentler, 1999). If model fit is insufficient, modification indices (MI) will be used to adjust the model within theoretically justifiable limits.

SECONDARY OUTCOMES:
Internal Consistency | Baseline
  Assessed using Cronbach's alpha coefficients for each factor. A value between 0.70 and 0.90 is considered to indicate appropriate internal consistency (Tavakol & Dennick, 2011).
Measurement Invariance | Baseline
  Evaluated using Multi-group CFA between office workers (VDT tasks) and production workers (physical tasks). Invariance is determined based on criteria such as ΔCFI ≤ 0.01 and ΔRMSEA ≤ 0.015 (Chen, 2007).
Construct Validity | Baseline
  Assessed by analyzing correlations (Pearson or Spearman) between the developed tool and standard instruments. A correlation coefficient (r) of ≥ 0.50 represents adequate convergent validity.
Cut-off Determination for Yellow Flags | Baseline
  Receiver Operating Characteristic (ROC) analysis will be conducted to establish optimal cut-off scores for identifying high-risk groups (Yellow flags). Established instruments (e.g., OSPRO-YF) will be used as a reference to calculate sensitivity, specificity, and the Youden index.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Biologics, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the privacy and confidentiality of the participants.